CLINICAL TRIAL: NCT00919191
Title: An Investigator-Blind, Phase 4 Study Assessing the Facial Irritation Potential of Two Acne Treatment Products Using A Split-Face Model
Brief Title: Evaluation of Irritation by Two Facial Gels Applied to Opposite Sides of the Face
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CA-P-6805
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: acne; irritation; objective sensory methods
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin; Adapalene; Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Two interventions in split-face model (Experimental): Once daily use in a split face model:
  1. Tretinoin gel
  2. Adapalene Benzoyl peroxide
  Interventions: Drug: Tretinoin gel; Drug: Adapalene and Benzoyl peroxide

INTERVENTIONS:
Drug: Tretinoin gel — Tretinoin gel 0.04% used once daily in a split-face model
  Other Names: Retin-A Micro Gel 0.04% Pump
Drug: Adapalene and Benzoyl peroxide — Adapalene .1% and Benzoyl peroxide 2.5%
  Other Names: Epiduo Gel

SUMMARY:
A study to compare the skin irritation potential of two marketed gels for acne treatment, each applied to half of the face of healthy volunteers.

DETAILED DESCRIPTION:
At the Baseline Visit, following satisfaction of entry criteria and screening procedures, all subjects will be applying two products to their faces, each on one side only. The side of the face receiving each product is randomly assigned. One group will use Retin-A MICRO Gel, (tretinoin) 0.04% Pump on the left side of the face and Epiduo Gel (adapalene .1% and benzoyl peroxide 2.5%), on the right side of the face daily for 3 consecutive weeks after washing with study-supplied facial wash. The other group will use the same products, but on opposite sides of the face for three consecutive weeks after washing with the same study-supplied facial wash.

Subjects will return to the study center every weekday morning for evaluation and application of both study products. Applications done on the weekends, will be done at home by the subject. At each visit the subject will be scored for cutaneous treatment effects by a blinded evaluator. At baseline and at the end of each week, subjects will be photographed and have chromometer readings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Before screening, subjects (or legally authorized representative) must read and sign the IRB approved Informed Consent Form (includes HIPPA and Photo release)
* Subjects must have Fitzpatrick Skin Type I, II or III, and judged by the Investigator to have healthy skin
* Subject's bilateral facial skin must be clear of any confounding irritation, rashes, acne, rosacea, etc. prior to the study
* Subject must be free of systemic retinoids for at least 2 months
* Subject must not be using any topical retinoids, systemic antibiotics, nicotinamide or systemic steroids for 1 month prior to study start
* All other topical medications to face (e.g., steroids, antimicrobials, salicylic acid and benzoyl peroxide) and cosmetics containing retinols, AHA's and bleaching agents such as hydroquinone are to be discontinued at least 2 weeks prior to study initiation
* Subjects will not apply any emollients and cosmetics to the facial area 24 hours prior to study initiation
* Subject must not be planning to become pregnant or nursing before entering the study and during the study period. In addition if using birth control pills, subject must be stabilized for at least 2 months. If subject is of child bearing potential, subject must be using approved method of birth control. Approved methods are birth control pills, implants, patches or spermicide with condoms.

Exclusion Criteria:

* Subjects who are pregnant or nursing
* Subjects who have a grade 1 or more for facial erythema
* Subjects who exhibit any skin condition (i.e., atopic dermatitis, seborrheic dermatitis, and psoriasis) or disease that may require concurrent therapy or may confound the evaluation of drug safety or efficacy
* Subjects who have a history of hypersensitivity to any of the formulation components listed in Appendix 1.
* Subjects who have received any experimental drug or used any experimental device 30 days prior to initiation of study therapy
* Subjects who have excessive facial hair that may obstruct or hinder the evaluation of any reactions
* Subjects who use any known photosensitizing agents
* Subjects who presently have skin cancer or actinic keratosis on the face

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rossi, MD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- Skin Study Center, Broomall, Pennsylvania, United States

REFERENCES:
- [Result] Leyden JJ, Nighland M, Rossi AB, Ramaswamy R. Irritation potential of tretinoin gel microsphere pump versus adapalene plus benzoyl peroxide gel. J Drugs Dermatol. 2010 Aug;9(8):998-1003. PMID 20684151
- See also: FDA's Drug Finder — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Tretinoin and Adapalene Benzoyl Peroxide Facial Gels: One group will use Retin-A MICRO Gel, (tretinoin) 0.04% Pump on the left side of the face and Epiduo Gel (adapalene .1% and benzoyl peroxide 2.5%), on the right side of the face daily for 3 consecutive weeks after washing with study-supplied facial wash. The other group will use the same products, but on opposite sides of the face for three consecutive weeks after washing with the same study-supplied facial wash.
Period: Overall Study
Arm/Group | Tretinoin and Adapalene Benzoyl Peroxide Facial Gels
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tretinoin and Adapalene Benzoyl Peroxide Facial Gels
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Comparative Assessment of Facial Irritation and Cutaneous Effects.
Description: Expert Grader Assessment, including cumulative scores for Erythema and Dryness on a scale of 0=none to 8=severe
Time Frame: Daily, for 3 weeks
Population: All participants used both gels concurrently, on opposite sides of the face (split-face model)
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Groups:
- Tretinoin Facial Gel: Tretinoin Facial Gel used once daily on one side of the face in a split face model
- Adapalene Benzoyl Peroxide Facial Gel: Adapalene Benzoyl Peroxide Facial Gel used once daily on the alternate side of the face in a split-face model
Arm/Group | Tretinoin Facial Gel | Adapalene Benzoyl Peroxide Facial Gel
Number analyzed (Participants) | 26 | 26
Scores on a Scale
  Cumulative Erythema | 1.1 (1.2) | 2.7 (7.8)
  Cumulative Dryness | 3.2 (5.3) | 6.2 (9.9)

2. Secondary Outcome: Self Assessment of Burning/Stinging and Itching
Description: Cumulative scores of Subjects' self assessment of burning/stinging and itching on a score from 0=none to 3=severe
Time Frame: Daily, for 3 weeks
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Groups:
- Tretinoin Facial Gel: Tretinoin Facial Gel used once daily on one side of the face in a split-face model
Arm/Group | Tretinoin Facial Gel | Adapalene Benzoyl Peroxide Facial Gel
Number analyzed (Participants) | 26 | 26
Scores on a Scale
  Cumulative Burning/Stinging | 1.4 (2.1) | 3.7 (4.8)
  Cumulative Itching | 0.7 (0.7) | 1.9 (3.0)

ADVERSE EVENTS:
Arm/Group | Tretinoin and Adapalene Benzoyl Peroxide Facial Gels
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less